CLINICAL TRIAL: NCT00190450
Title: Multicentric Intracerebral Grafting in Huntington's Disease
Brief Title: MIG-HD: Multicentric Intracerebral Grafting in Huntington's Disease
Acronym: MIG-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 001106
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Huntington Disease
Keywords: Huntington; graft; cellular therapy; striatum
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Early Graft (Early G)
  Interventions: Biological: graft intracerebral of foetal neurons
- 2 (Experimental): Late Graft (Late G)
  Interventions: Biological: graft intracerebral of foetal neurons

INTERVENTIONS:
Biological: graft intracerebral of foetal neurons — graft intracerebral of foetal neurons

SUMMARY:
The aim of this study is to assess the clinical benefit of intrastriatal grafting of human cells from the foetal ganglionic eminence in patients with Huntington's disease. The duration of the study will be 52 months. A first group of patients will be grafted at M13-14 (early G group) and a second group of patients will be grafted at M33-34 (late G group). The principal criterion is the comparison of the progression between M12 and M32 of the motor score (TMS) of the UHDRS between grafted patients (early G group) and not yet grafted patients (late G group). An additional evaluation will be performed to compare the progression in individual patients over the 52-month study period. We will thus be able to compare the pre and post-graft TMS progression for all patients.

DETAILED DESCRIPTION:
The aim of this study is to show the existence of a clinical benefit rising from a substitution of the striatal neurons degenerated among a large cohort of Huntington's patient at early stage by homologous neurons coming from human foetuses, This effect will be estimated, compared with a group of patients not treated at first, on the results of the motor scale of the Unified Huntington Disease Rating Scale (UHDRS, Huntington study group, on 1996).

Transplants will be realized in two surgical times to avoid the risk of hurts per-operating, BI-CAUDES, if transplants were realized at single time. The minimal interval between both transplants will be of 2 weeks, so as to let the patient recover of the first general anaesthesia It's a multicentric study of phase II randomised and controlled, with direct individual benefit.

ELIGIBILITY:
Inclusion Criteria:

* Disease clinically declared since at least 1 year ,UHDRS motor > or =5
* TFC > or = 10.
* CAG > or = 36
* Age between 18 and 65
* Family and socially integrated subject
* Informed consent.

Exclusion Criteria:

* Severe intellectual deterioration or neuropsychiatric disorders making the follow-up longitudinal too complicated (score MATTIS < 120).
* Not-observance of the appointments and the symptomatic treatments in pre-surgical period.
* Intercurrent disease making a surgical operation impossible.
* Associated disease having a neurological repercussion, intercurrent cerebral lesion with the IRM.
* Visceral affection engraves, evolutionary, which brings into play the vital forecast or makes risks for general anaesthesia.
* Mental Affection likely to disturb adhesion with the protocol, and in particular antecedents of hallucinations spontaneous and/or induced by the drugs; antecedents of serious depression having required repeated hospitalizations; antecedents of repeated suicide attempts.
* Cerebral morphological anomalies, others that those characteristic of the disease, noted with the IRM or the tomodensitometry.
* Participation in progress, or stopped since less than three months, with a therapeutic protocol of the Huntington's disease Exclusion Criteria (pre-randomization)
* TFC < 8
* Not-observance of the appointments and the symptomatic treatments in pre-surgical period.
* Intercurrent disease returning the surgery or impossible immunosuppression. v Subject completely isolated with his family and socially..
* UHDRS motor < 5.
* Positives serologies for HIV1, HIV2, AgP24, HTLV1 et 2, HEPATITE B, HEPATITE C, syphilis
* Psychiatric disorders being able to compromise the follow-up.
* Signs other than Huntington with the IRM.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2002-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Motor UHDRS rating scale, at randomization, 20 month after transplant | during de study

SECONDARY OUTCOMES:
Neurologic, Cognitive, Neurophysiologic, Psychiatric, MRI and Pet-scan evaluation at randomization, 20 month after and at the end of the protocol | during the study

CONTACTS AND LOCATIONS:
Overall Officials: A-C. BACHOUD-LEVI, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Henri Mondor, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Bachoud-Levi AC, Remy P, Nguyen JP, Brugieres P, Lefaucheur JP, Bourdet C, Baudic S, Gaura V, Maison P, Haddad B, Boisse MF, Grandmougin T, Jeny R, Bartolomeo P, Dalla Barba G, Degos JD, Lisovoski F, Ergis AM, Pailhous E, Cesaro P, Hantraye P, Peschanski M. Motor and cognitive improvements in patients with Huntington's disease after neural transplantation. Lancet. 2000 Dec 9;356(9246):1975-9. doi: 10.1016/s0140-6736(00)03310-9. PMID 11130527
- [Derived] Kinfe T, Del Vecchio A, Nussel M, Zhao Y, Stadlbauer A, Buchfelder M. Deep brain stimulation and stereotactic-assisted brain graft injection targeting fronto-striatal circuits for Huntington's disease: an update. Expert Rev Neurother. 2022 Sep;22(9):781-788. doi: 10.1080/14737175.2022.2091988. Epub 2022 Jun 29. PMID 35766355
- [Derived] Riad R, Lunven M, Titeux H, Cao XN, Hamet Bagnou J, Lemoine L, Montillot J, Sliwinski A, Youssov K, Cleret de Langavant L, Dupoux E, Bachoud-Levi AC. Predicting clinical scores in Huntington's disease: a lightweight speech test. J Neurol. 2022 Sep;269(9):5008-5021. doi: 10.1007/s00415-022-11148-1. Epub 2022 May 14. PMID 35567614
- [Derived] Bachoud-Levi AC; on behalf the Multicentric Intracerebral Grafting in Huntington's Disease Group. Human Fetal Cell Therapy in Huntington's Disease: A Randomized, Multicenter, Phase II Trial. Mov Disord. 2020 Aug;35(8):1323-1335. doi: 10.1002/mds.28201. Epub 2020 Jul 15. PMID 32666599
- [Derived] Schramm C, Katsahian S, Youssov K, Demonet JF, Krystkowiak P, Supiot F, Verny C, Cleret de Langavant L, Bachoud-Levi AC; European Huntington's Disease Initiative Study Group and the Multicentre Intracerebral Grafting in Huntington's Disease Group. How to Capitalize on the Retest Effect in Future Trials on Huntington's Disease. PLoS One. 2015 Dec 29;10(12):e0145842. doi: 10.1371/journal.pone.0145842. eCollection 2015. PMID 26714284
- [Derived] Teichmann M, Gaura V, Demonet JF, Supiot F, Delliaux M, Verny C, Renou P, Remy P, Bachoud-Levi AC. Language processing within the striatum: evidence from a PET correlation study in Huntington's disease. Brain. 2008 Apr;131(Pt 4):1046-56. doi: 10.1093/brain/awn036. Epub 2008 Mar 11. PMID 18334537
- See also: Huntington french speaking network website — http://www.hdnetwork.org/